CLINICAL TRIAL: NCT02008214
Title: Efficacy of Pentoxyfylline Addition to a Treatment Scheme Based on Interferon Alpha and Ribavirin on Hepatitis C Virus Coinfected HIV Patients, Considering Interleukin 28B Polymorphism rs12979860
Brief Title: Efficacy of PTX+IFN Alpha+ RBV on Hepatitis C Virus Coinfected HIV Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, JAIME ANDRADE VILLANUEVA, Professor-Investigator, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTX-HCV/HIV
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Hepacivirus; HIV Infections
Keywords: Pentoxifylline; Sustained virologic response; Hepatic fibrosis
MeSH Terms: conditions — HIV Infections; Liver Cirrhosis | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTX (Experimental): IFN 180 micrograms subcutaneous weekly RBV 400 mg each 12 h, oral PTX 400 mg each 12 h, oral
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): IFN 180 micrograms subcutaneous weekly RBV 400 mg each 12 h, oral Placebo oral daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Addition of pentoxifylline to current HCV treatment
  Arms: PTX
Drug: Placebo — Placebo matching pentoxifylline dosage
  Arms: Placebo

SUMMARY:
Current Hepatitis C virus (HCV) treatment consists of the combination of interferon alpha 2a (IFN-alpha 2a) plus ribavirin (RBV) and it provides sustained virologic responses (SVR) on 54 to 56% on HCV monoinfected patients and this response is even lower on HIV-HCV coinfected patients. A previous study on HCV monoinfected patients showed that the addition of pentoxyfylline (PTX) to a treatment scheme based on interferon-alfa and ribavirin increased SVR on 25%, although it is not known if the same effect is to be obtained in HCV-HIV coinfected patients.

On the other hand, other factors such as host genetics, have proved to influence treatment response on HCV infected patients. The best described genetic factor so far is the interleukin 28B (IL28B) polymorphism rs12979860, where a cytosine-cytosine (CC) genotype provides an almost twice increase on SVR than the rest of the genotypes.

Therefore, this is a randomized, double blind study to assess the efficacy of pentoxyfylline addition to a treatment scheme based on interferon-alfa and ribavirin in chronic HCV genotype 1, co-infected HIV-1 positive subjects, considering the IL28B polymorphism rs12979860.

HIV-HCV coinfected subjects currently receiving Highly active antiretroviral therapy (HAART), with at least 8 months on undetectable HIV viral load and T helper cells count of 200 or higher will be included. Patients will be randomized on one of two groups:

* Group A: IFN alpha 2a + RBV + PTX
* Group B: IFN alpha 2a + RBV + placebo

Patients will be followed for primary outcome during 72 (for rapid responders) or 96 weeks (for non rapid responses). Outcome measures will be the following:

* SVR rate 24 weeks after the end of treatment
* Grade of Hepatic fibrosis from baseline to the end of treatment, measured by transient elastography and the AST to platelet ratio index (APRI index)
* IL28B rs12979860 genotype

The study hypothesis is that the addition of PTX to a treatment scheme based on IFN-alfa2a and RBV in chronic HCV genotype 1, co-infected HIV-1 positive subjects will improve SVR rate and fibrosis progression irrespectively of IL28B rs12979860 genotype.

ELIGIBILITY:
Inclusion Criteria:

* HIV/HCV coinfected patients
* 18 to 65 years old
* currently receiving HAART
* non-pregnant women
* HIV infection controlled as: undetectable viral load (<40 copies/mL) for at least 8 months and T helper cells count of 200 cells/μL or above
* no contraindications to IFN alpha2a, RBV or PTX treatment
* sign informed consent form
* laboratory parameters within acceptable ranges

Exclusion Criteria:

* Women that present a positive pregnancy test during the study
* Patients that for any reason no longer wish to receive IFN alpha2a, RBV or PTX treatment
* Serious adverse events that prevent to continue IFN alpha2a, RBV or PTX treatment; such as severe neutropenia, severe thrombocytopenia or severe anemia
* Presence of an opportunistic infection or malignancy that requires treatment with drugs interacting with IFN alpha2a, RBV or PTX
* Patients that fail to adhere to treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
sustained virologic rate 24 weeks post treatment with IFNalpha 2a/RBV/PTX with genotype 1 chronic HCV infection + HIV infection | SVR rate at 24 weeks after the end of therapy
  Primary objective: is to evaluate sustained virologic response at post treatment week 24 following treatment with IFNalpha 2a/RBV/PTX with genotype 1 chronic HCV infection + HIV infection

SECONDARY OUTCOMES:
grade of hepatic fibrosis | Baseline and week 72 (for quick responders) or week 96 (for non-quick responders)
  The liver stiffness (hepatic fibrosis) will be measured by transient elastography and the APRI index on the baseline visit and then at the follow up visit after treatment, which will be after 72 weeks, for patients that turn out to be quick responders; or 96 weeks, for patients that turn out to be non-quick responders.
rapid virologic response (RVR) and extended rapid virologic response (eRVR) rates | RVR at week 4 and eRVR at week 48 post treatment
  secondary objective (2): Evaluate rapid virologic response (RVR) and extended rapid virologic response (eRVR)

OTHER OUTCOMES:
Percentage of patients with CC genotype on the IL28B rs12979860 polymorphism | week 72
  We will compare the percentage of patients with CC genotype among patients that achieved sustained virologic response and those who did not achieved it. This is to confirm if the intervention provides a beneficial effect, irrespectively of host genetic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil de Guadalajara, Guadalajara, Jalisco, Mexico